CLINICAL TRIAL: NCT05376891
Title: Disease Registry on Patients With Advanced NSCLC Harboring METex14 Skipping Alterations (MOMENT)
Brief Title: Met Non Small Cell Cancer Registry (MOMENT)
Status: Recruiting | Type: Observational
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Other Study IDs: MS200095_0050
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Cancer
Keywords: Disease Registry; METex14 Skipping Alterations
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Advanced Non-small Cell Lung Cancer with METex14 skipping alterations: Participants diagnosed with advanced NSCLC and who receive available therapies in routine clinical practice setting will be part of this registry. Data will be collected routinely from the point of enrollment of a participants into the registry until death, loss to follow-up (drop-out), subsequent enrollment into a clinical trial, or end of data collection period for the registry.

SUMMARY:
The purpose of this multi-national disease registry is to collect prospectively (with longitudinal follow-up) high-quality, standardized, and contemporaneous data to capture changes in the non-small cell lung cancer (NSCLC) treatment landscape and outcomes over time.

The registry will capture data on participants; demographic, clinical characteristics (including biomarker data), treatment patterns, and effectiveness and safety outcomes for advanced NSCLC with mesenchymal-epithelial transition exon 14 (METex14) participants treated with systemic therapy.

DETAILED DESCRIPTION:
This is a disease registry, which is an organized system using non-interventional methods to collect data on a patient population defined by a particular disease, exposure, or condition, and which is followed over time. Non-interventional means that after participants enrollment, participants will be treated according to the routine clinical treatment decision by the physician. The registry will not impose any treatment or procedure for participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants who signed ICF
* Participants with advanced stage (stages IIIB-IV) NSCLC (all histologies) and Confirmed METex14 skipping alterations (by valid assay)
* Participants who are starting or are already being treated with systemic therapy

Exclusion Criteria:

* Participants who are enrolled in a clinical trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with advanced stage (stages IIIB-IV) NSCLC and confirmed METex14 skipping alterations who are initiating or already treated with a systemic therapy will be included.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2022-10-04 (Actual); Primary Completion 2028-04-28 (Estimated); Study Completion 2028-04-28 (Estimated)

PRIMARY OUTCOMES:
Best Overall Response (BOR) | Through study completion, up to approximately 4.9 years
Tumor Response According to Response Evaluation Criteria in Solid Tumors Version (RECIST) 1.1 | Up to approximately 4.9 years
Overall Survival (OS) | Through study completion, up to approximately 4.9 years
Number of Participants with Adverse Events (AEs) | Up to approximately 4.9 years
Number of Participants with Adverse Reactions (ARs) | Up to approximately 4.9 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (60):
- United States (3):
  - Holy Cross Health, Fort Lauderdale, Florida
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Austria (2):
  - Klinikum Klagenfurt Am Woerthersee, Klagenfurt
  - Klinik Floridsdorf, Vienna
- Belgium (2):
  - AZ Delta, Roeselare
  - AZ Nikolaas, Sint-Niklaas
- Canada (2):
  - Ottawa Hospital General Campus, Ottawa
  - Princess Margaret Cancer Centre, Toronto
- Czechia (2):
  - FN Olomouc, Olomouc
  - University Hospital Na Bulovce, Prague
- France (7):
  - Centre Hospitalier de Cholet, Cholet
  - CHRU Lille, Lille
  - Hôpital du Scorff, Lorient
  - Centre Leon Berard, Lyon
  - Hospital Tenon & University Paris 6, Paris
  - Institut Curie - Centre de Lutte Contre le Cancer (CLCC), Paris
  - CHU de Toulouse Hopital Larrey, Toulouse
- Germany (4):
  - Klinikum Chemnitz GmbH, Chemnitz
  - KKH Grosshansdorf GmbH, Großhansdorf
  - Thoraxklinik-Heidelberg gGmbH, Heidelberg
  - Klinik Löwenstein GmbH, Löwenstein
- Israel (8):
  - Haemek Medical Center, Afula
  - Bnei-Zion Medical Center, Haifa
  - Carmel Medical Center, Haifa
  - Rambam Medical Center - PPDS, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Rabin Medical Center Oncology Beilinson Campus, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (6):
  - Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale Dei Tumori, Milan
  - AOU dell'Università degli Studi della Campania Luigi Vanvitelli, Napoli
  - I.F.O. Istituto Nazionale Tumori Regina Elena IRCCS, Rome
  - Azienda Sanitaria Ospedaliera S Luigi Gonzaga, Torino
  - Ospedale di Circolo, Varese
- Netherlands (3):
  - VU Medisch Centrum, Amsterdam
  - Universitair Medisch Centrum Groningen - Department of Medical Oncology, Groningen
  - Leiden University Medical Center, Leiden
- Portugal (3):
  - Centro Hospitalar de Lisboa Norte, EPE - Hospital de Santa Maria, Lisbon
  - Centro Hospitalar do Porto E.P.E. Hospital de Santo António, Porto
  - Instituto Portugues de Oncologia Do Porto Francisco Gentil Epe - PPDS, Porto Covo
- Spain (9):
  - Clinica Tres Torres, Barcelona
  - Institut Universitari Dexeus-Quiron - Servei d oncologia medica - Institut Oncologic Dr. Rosell, Barcelona
  - Complejo Hospitalario Universitario Insular-Materno Infantil, Las Palmas de Gran Canaria
  - Centro Integral Oncologico Clara Campa, Madrid
  - Centro Oncologico MD Anderson, Madrid
  - Hospital Regional Universitario de Malaga - Hospital General, Málaga
  - Hospidal Universitario Ntra. Sra. De Valme, Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Universitetssjukhuset i Linköping, Linköping, Sweden
- United Kingdom (8):
  - Bedford General Hospital, Bedford
  - Birmingham Heartlands Hospital, Birmingham
  - Royal Bournemouth Hospital, Bournemouth
  - The Royal Marsden Hospital, Chelsea
  - Northwick Park Hospital, Harrow
  - Clatterbridge Cancer Centre - Liverpool, Liverpool
  - Charing Cross Hospital, London
  - Preston Hospital, Preston

REFERENCES:
- [Derived] Thomas M, Christopoulos P, Iams WT, Mazieres J, Cortot AB, Peled N, Minuti G, Smit EF, Audhuy F, Berghoff K, Eggleton SP, Fries F, Hildenbrand M, Liu P, Mahmoudpour SH, Menzel C, Oksen D. MOMENT registry: Patients with advanced non-small-cell lung cancer harboring MET exon 14 skipping treated with systemic therapy. J Comp Eff Res. 2025 Feb;14(2):e240127. doi: 10.57264/cer-2024-0127. Epub 2025 Jan 21. PMID 39836056
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200095_0050
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html